CLINICAL TRIAL: NCT02759224
Title: A Study to Compare the Pharmacokinetics of Lafutidine and Irsogladine Maleate Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-LIC-CT-101
Record Dates: First submitted 2016-04-21; First posted 2016-05-03 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — lafutidine; irsogladine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Lafutidine and Irsogladine maleate --> BRI-1501) (Other): Subjects of Arm A take Lafutidine and Irsogladine maleate Individual tablets at 1st day as period I. And then, after wash out for 35 days, as period II, subjects of Arm A take a BRI-1501 tablet at 36th day
  Interventions: Drug: BRI-1501; Drug: Lafutidine; Drug: Irsogladine maleate
- Arm B (BRI-1501 --> Lafutidine and Irsogladine maleate) (Other): Subjects of Arm B take a BRI-1501 tablet at 1st day as period I. And then, after wash out for 35 days, as period II, subjects of Arm B take Lafutidine and Irsogladine maleate Individual tablets at 36th day
  Interventions: Drug: BRI-1501; Drug: Lafutidine; Drug: Irsogladine maleate

INTERVENTIONS:
Drug: BRI-1501
Drug: Lafutidine
Drug: Irsogladine maleate

SUMMARY:
An Open-Label, Randomized, Single-dose, 2x2 Crossover Study to Compare the Pharmacokinetics of BRI-1501 Tablet and Coadministration of Lafutidine and Irsogladine maleate as Individual Tablets in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, aged 19- 50 years

Exclusion Criteria:

* History of clinically significant and active disease
* History of gastrointestinal disease
* History of clinically significant hypersensitivity to study drug, any other drug
* Laboratory test serum AST or ALT > 1.25 times of upper normal range serum total bilirubin > 1.5 times of upper normal range eGFR < 60 ml/min/1.73m² serological test(HBsAg, HCV Ab, HIV Ag/Ab, Syphilis reagin) positive
* Hypotension or hypertension
* Pregnant or nursing women
* Participation in any other study within 90 days

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration(Cmax) of Lafutidine and Irsogladine maleate | 0~36 hour after medication
Area under the plasma drug concentration-time curve(AUClast) of Lafutidine and Irsogladine maleate | 0~36 hour after medication

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, South Korea